CLINICAL TRIAL: NCT01083433
Title: Intensive Diabetes Clinic and Intermittent Continuous Glucose Monitoring in Adolescents With Type 1 Diabetes Mellitus in Poor Glycemic Control
Brief Title: Study to Find Out if Intensive Diabetes Clinic and Continuous Glucose Monitors Help Teenagers With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sarah A. MacLeish, Physician, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBCDM-01; MH018830 (Other Grant/Funding Number: TRN503976)
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Results first posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Continuous Glucose Monitor; Adherence; Adolescents; Diabetes Education
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Diabetes Care (No Intervention): Patients will attend diabetes clinic as usual, once every 3 months.
- Intensive Diabetes Clinic (Experimental): Patients will attend diabetes clinic on a monthly basis for 4 months in a row. Each patient will have a 30 minute visit with a physician, 30 minutes dedicated to diabetes education, and 45 minutes with a child psychologist.
  Interventions: Behavioral: Diabetes related psychological counseling and education
- Intensive Diabetes Clinic plus CGM (Experimental): Patients in this group will include all procedures as listed for group 2 (intensive diabetes clinic) in addition to wearing a continuous glucose monitor for 3-5 days each month. Patients will also have an additional 30 minutes with a psychology graduate student dedicated to adherence with the CGM.
  Interventions: Behavioral: Diabetes related psychological counseling and education; Device: Continuous Glucose Monitor

INTERVENTIONS:
Behavioral: Diabetes related psychological counseling and education — The psychology intervention is based in part on an intervention to maintain parental support for diabetes care in adolescence which was developed by Anderson and colleagues (1999). The first session will include education to parents and children regarding the importance of sharing responsibility for treatment related tasks. The second session will include a discussion of the treatment sharing plan developed at the first visit and problems that may have occurred will be discussed. The third session will include a discussion of planning for possible future problems. Visits 1, 2, and 3 will include 30 minutes of diabetes education.
  Other Names: Diabetes Education; Diabetes Psychological Counseling
  Arms: Intensive Diabetes Clinic; Intensive Diabetes Clinic plus CGM
Device: Continuous Glucose Monitor — Patients in the intensive diabetes clinic plus CGM group will wear the iPro after the baseline visit followed by every month for 4 months.
  Other Names: Medtronic Minimed iPro
  Arms: Intensive Diabetes Clinic plus CGM

SUMMARY:
The purpose of this research study is to find out ways to help pre-teens and teens and their families to improve diabetes control and to help with the burden of diabetes management. Specifically, the study aims to find out if coming to diabetes clinic more frequently and for a longer period of time helps adolescents with diabetes, and if adolescents who wear a continuous glucose monitor (CGM) for 3-5 days a month will have better diabetes control.

DETAILED DESCRIPTION:
Good glycemic control is critical in preventing chronic complications of type 1 diabetes. However, achieving good glycemic control remains elusive for many adolescents. This study evaluates two clinic-based approaches for improving glycemic control in adolescents with poorly controlled type 1 diabetes - an intensive diabetes support and education program alone and the same intensive diabetes support and education program together with continuous glucose monitoring - in comparison with standard diabetes care.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus of at least 12 months duration, followed by Rainbow Babies and Children's Pediatric Endocrinology and Diabetes Division
* Most recent HbA1c >= 8.5%
* Patients must be willing to check their blood sugar at least 4 times daily while wearing the CGM
* Patients and families must be willing to come to diabetes clinic once a month for 4 months

Exclusion Criteria:

* Inability to understand and/or speak the English language
* Pregnancy
* Psychological counseling with Dr. Rebecca Hazen regarding diabetes adherence prior to the study

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A MacLeish, D.O., Principal Investigator — UHCMC Division of Pediatric Endocrinology; Rebecca A Hazen, Ph.D., Principal Investigator — UHCMC Division of Behavioral Pediatrics; Leona Cuttler, M.D, Principal Investigator — UHCMC Division of Pediatric Endocrinology; Rose Gubitosi-Klug, M.D, Ph.D., Principal Investigator — UHCMC Division of Pediatric Endocrinology
Locations (1):
- UHCMC, Cleveland, Ohio, United States

REFERENCES:
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Monnier L, Mas E, Ginet C, Michel F, Villon L, Cristol JP, Colette C. Activation of oxidative stress by acute glucose fluctuations compared with sustained chronic hyperglycemia in patients with type 2 diabetes. JAMA. 2006 Apr 12;295(14):1681-7. doi: 10.1001/jama.295.14.1681. PMID 16609090
- [Background] Monnier L, Colette C. Glycemic variability: should we and can we prevent it? Diabetes Care. 2008 Feb;31 Suppl 2:S150-4. doi: 10.2337/dc08-s241. PMID 18227477
- [Background] Weber C, Schnell O. The assessment of glycemic variability and its impact on diabetes-related complications: an overview. Diabetes Technol Ther. 2009 Oct;11(10):623-33. doi: 10.1089/dia.2009.0043. PMID 19821754
- [Background] El-Osta A, Brasacchio D, Yao D, Pocai A, Jones PL, Roeder RG, Cooper ME, Brownlee M. Transient high glucose causes persistent epigenetic changes and altered gene expression during subsequent normoglycemia. J Exp Med. 2008 Sep 29;205(10):2409-17. doi: 10.1084/jem.20081188. Epub 2008 Sep 22. PMID 18809715
- [Background] Hirsch IB. Glycemic variability: it's not just about A1C anymore! Diabetes Technol Ther. 2005 Oct;7(5):780-3. doi: 10.1089/dia.2005.7.780. No abstract available. PMID 16241882
- [Background] Monnier L, Colette C, Owens DR. Glycemic variability: the third component of the dysglycemia in diabetes. Is it important? How to measure it? J Diabetes Sci Technol. 2008 Nov;2(6):1094-100. doi: 10.1177/193229680800200618. PMID 19885298
- [Background] Deiss D, Bolinder J, Riveline JP, Battelino T, Bosi E, Tubiana-Rufi N, Kerr D, Phillip M. Improved glycemic control in poorly controlled patients with type 1 diabetes using real-time continuous glucose monitoring. Diabetes Care. 2006 Dec;29(12):2730-2. doi: 10.2337/dc06-1134. No abstract available. PMID 17130215
- [Background] Schaepelynck-Belicar P, Vague P, Simonin G, Lassmann-Vague V. Improved metabolic control in diabetic adolescents using the continuous glucose monitoring system (CGMS). Diabetes Metab. 2003 Dec;29(6):608-12. doi: 10.1016/s1262-3636(07)70076-9. PMID 14707890
- [Background] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Tamborlane WV, Beck RW, Bode BW, Buckingham B, Chase HP, Clemons R, Fiallo-Scharer R, Fox LA, Gilliam LK, Hirsch IB, Huang ES, Kollman C, Kowalski AJ, Laffel L, Lawrence JM, Lee J, Mauras N, O'Grady M, Ruedy KJ, Tansey M, Tsalikian E, Weinzimer S, Wilson DM, Wolpert H, Wysocki T, Xing D. Continuous glucose monitoring and intensive treatment of type 1 diabetes. N Engl J Med. 2008 Oct 2;359(14):1464-76. doi: 10.1056/NEJMoa0805017. Epub 2008 Sep 8. PMID 18779236

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensive Diabetes Clinic Plus CGM: Patients in this group will include all procedures as listed for group 2 (intensive diabetes clinic) in addition to wearing a CGM for 3-5 days each month. Patients will also have an additional 30 minutes with a psychology graduate student dedicated to adherence with the CGM.
  Diabetes related psychological counseling and education: The psychology intervention is based in part on an intervention to maintain parental support for diabetes care in adolescence which was developed by Anderson and colleagues (1999). The first session will include education to parents and children regarding the importance of sharing responsibility for treatment related tasks. The second session will include a discussion of the treatment sharing plan developed at the first visit and problems that may have occurred will be discussed. The third session will include a discussion of planning for possible future problems. Visits 1, 2, and 3 will include 30 minutes of diabetes education.
Period: Overall Study
Arm/Group | Standard Diabetes Care | Intensive Diabetes Clinic | Intensive Diabetes Clinic Plus CGM
Started | 22 | 23 | 23
Completed | 20 | 17 | 18
Not Completed | 2 | 6 | 5
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 5 | 3
Not completed — Pregnancy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intensive Diabetes Clinic Plus CGM: Patients in this group will include all procedures as listed for group 2 (intensive diabetes clinic) in addition to wearing a continuous glucose monitor for 3-5 days each month. Patients will also have an additional 30 minutes with a psychology graduate student dedicated to adherence with the CGM.
  Diabetes related psychological counseling and education: The first session will include education to parents and children regarding the importance of sharing responsibility for treatment related tasks. The second session will include a discussion of the treatment sharing plan developed at the first visit and problems that may have occurred will be discussed. The third session will include a discussion of planning for possible future problems. Visits 1, 2, and 3 will include 30 minutes of diabetes education.
  Continuous Glucose Monitor: Patients in the intensive diabetes clinic plus CGM group will wear the iPro after the baseline visit followed by every month for 4 months.
- Total: Total of all reporting groups
Arm/Group | Standard Diabetes Care | Intensive Diabetes Clinic | Intensive Diabetes Clinic Plus CGM | Total
Number analyzed (Participants) | 22 | 23 | 23 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (2.6) | 14.9 (2.6) | 14.6 (2.2) | 14.6 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 15 | 42
  Male | 8 | 10 | 8 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 6 | 17
  White | 14 | 15 | 16 | 45
  More than one race | 2 | 3 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
HbA1c [Mean (Standard Deviation); unit: percent] | 11.0 (2.2) | 9.9 (1.3) | 10.0 (1.4) | 10.3 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control
Description: Serum hemoglobin A1c (HbA1c) will be measured in all groups at the baseline visit and visit 4.
Time Frame: Baseline and visit 4
Measure: Mean (Standard Deviation); unit: percent HbA1c
Arm/Group | Standard Diabetes Care | Intensive Diabetes Clinic | Intensive Diabetes Clinic Plus CGM
Number analyzed (Participants) | 20 | 17 | 18
percent HbA1c
  VISIT 4 | 10.8 (2.2) | 9.43 (1.1) | 9.4 (0.9)
  BASELINE | 11.0 (2.1) | 9.93 (1.3) | 10.0 (1.4)

2. Secondary Outcome: Insulin Dose Changes
Description: Insulin doses in units per kilogram per day will be calculated at baseline and visit 4.
Time Frame: Baseline and visit 4
Measure: Mean (Standard Deviation); unit: u/kg/day
Arm/Group | Standard Diabetes Care | Intensive Diabetes Clinic | Intensive Diabetes Clinic Plus CGM
Number analyzed (Participants) | 20 | 17 | 18
u/kg/day
  VISIT 4 | 1.02 (0.3) | 1.03 (0.3) | 1.10 (0.3)
  BASELINE | 0.98 (0.3) | 1.09 (0.4) | 1.0 (0.3)

3. Secondary Outcome: Number of Hypoglycemic Excursions (CGM Glucose <70 mg/dL)
Description: CGM downloads at baseline and visit 4 will be used to tabulate the number of episodes of blood glucoses < 70 mg/dL. At each visit patients will be asked to recall any episodes of severe hypoglycemia that occurred since the last visit. Data from the continuous glucose monitors will be used to evaluate the percent of time that patients are below 70 mg/dL and the number of glucose excursions below 70 mg/dL. Total number of excursions under 70 mg/dL from baseline to visit 4 will be added together.
Time Frame: Total from baseline to visit 4
Measure: Mean (Standard Deviation); unit: number of hypoglycemic excursions
Groups:
- Intensive Diabetes Clinic Plus CGM: Patients in this group will include all procedures as listed for group 2 (intensive diabetes clinic) in addition to wearing a continuous glucose monitor for 3-5 days each month. Patients will also have an additional 30 minutes with a psychology graduate student dedicated to adherence with the CGM.
  Diabetes related psychological counseling and education: Same as Intensive diabetes clinic group.
  Continuous Glucose Monitor: Patients in the intensive diabetes clinic plus CGM group will wear the iPro after the baseline visit followed by every month for 4 months.
Arm/Group | Standard Diabetes Care | Intensive Diabetes Clinic | Intensive Diabetes Clinic Plus CGM
Number analyzed (Participants) | 22 | 23 | 23
number of hypoglycemic excursions
  Baseline | 3.3 (3.3) | 3.7 (3.3) | 3.8 (3.8)
  Visit 4 | 2.9 (2.0) | 4.4 (3.8) | 4.0 (5.3)

4. Secondary Outcome: Adherence to Prescribed Diabetes Regimen
Description: Diabetes Self Management Profile, given to participant (child) at baseline and visit 4. Minimum score zero, maximum score 88. A higher score indicates better adherence. The DSMP is a 10-15 minute, 25-question, validated, structured interview of adherence with diabetes self-management tasks administered separately to parents and youth. It was verbally administered by one pediatric endocrinologist and one trained research assistant. It assesses self-management of exercise and hypoglycemia (7 questions), carbohydrate counting and insulin dose calculation (6 questions), blood glucose and ketone monitoring (8 questions), and insulin timing and dosing (4 questions).
Time Frame: Baseline and visit 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Standard Diabetes Care | Intensive Diabetes Clinic | Intensive Diabetes Clinic Plus CGM
Number analyzed (Participants) | 20 | 17 | 18
Score on a scale
  VISIT 4 | 51 (12.4) | 58.0 (8.7) | 54.9 (8.9)
  BASELINE | 47.3 (10.6) | 50.2 (11.2) | 50.9 (9.8)

5. Secondary Outcome: Satisfaction With Intensive Diabetes Clinic and Usage of the Continuous Glucose Monitor
Description: Survey of patient and parent satisfaction in the interventions groups only, satisfaction with the overall study including CGM use and psychological intervention. Satisfaction measured on a 7 point Likert scale, with highest satisfaction at a score of 7 and lowest score 1.
Time Frame: Visit 4
Population: Some parents did not fill out the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intensive Diabetes Clinic | Intensive Diabetes Clinic Plus CGM
Number analyzed (Participants) | 17 | 18
score on a scale
  Overall Patient Satisfaction | 6.3 (0.8) | 5.5 (1.4)
  Overall Parent Satisfaction: number analyzed (Participants) | 14 | 16
  Overall Parent Satisfaction | 6.1 (1.1) | 6.6 (0.6)

6. Secondary Outcome: Diabetes Knowledge
Description: The Diabetes Knowledge Questionnaire was adapted from Butler et al. It is a written questionnaire, self administered independently to parents and children to assess their knowledge about diabetes management. It includes 37 multiple choice questions assessing basic information about diabetes, how to deal with diabetes-related tasks, and management of hypothetical situations. A total score out of 37 possible points is computed for diabetes knowledge, score can range from 0-37. A higher score indicates higher knowledge.
Time Frame: Baseline and month 4
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intensive Diabetes Clinic Plus CGM: Patients in this group will include all procedures as listed for group 2 (intensive diabetes clinic) in addition to wearing a continuous glucose monitor for 3-5 days each month. Patients will also have an additional 30 minutes with a psychology graduate student dedicated to adherence with the CGM.
  Diabetes related psychological counseling and education: same as description for intensive diabetes clinic group.
  Continuous Glucose Monitor: Patients in the intensive diabetes clinic plus CGM group will wear the iPro after the baseline visit followed by every month for 4 months.
Arm/Group | Standard Diabetes Care | Intensive Diabetes Clinic | Intensive Diabetes Clinic Plus CGM
Number analyzed (Participants) | 20 | 17 | 18
score on a scale
  Parents baseline knowledge | 33 (3.3) | 33 (2.0) | 31 (3.9)
  Parents visit 4 | 33 (2.1) | 33 (2.3) | 33 (2.4)
  Patients baseline | 27 (5.9) | 28 (7.7) | 26 (5.8)
  Patients visit 4 knowledge | 29 (5.4) | 29 (9.1) | 29 (4.7)

ADVERSE EVENTS:
Arm/Group | Standard Diabetes Care | Intensive Diabetes Clinic | Intensive Diabetes Clinic Plus CGM
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 4/22 | 1/23 | 2/23
Other Adverse Events (participants affected / at risk) | 1/22 | 0/23 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Diabetes Care (N=22) | Intensive Diabetes Clinic (N=23) | Intensive Diabetes Clinic Plus CGM (N=23)
Diabetic Ketoacidosis (Endocrine disorders) | 4 (5) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Diabetes Care (N=22) | Intensive Diabetes Clinic (N=23) | Intensive Diabetes Clinic Plus CGM (N=23)
Continuous Glucose Monitor Site Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Minor site infection requiring topical antibiotics.

LIMITATIONS AND CAVEATS:
* High rate of attrition and lack of outcome data in patients lost to follow-up.
* Lack of CGM alone group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No